CLINICAL TRIAL: NCT02407730
Title: EFFects of Thrombophilia on the Outcomes of Assisted Reproduction
Brief Title: EFFects of Thrombophilia on the Outcomes of Assisted Reproduction Technologies
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Marcello Di Nisio, Principal Investigator, G. d'Annunzio University
Other Study IDs: EFFORT
Record Dates: First submitted 2015-03-20; First posted 2015-04-03 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Birth Rate; Embryo Implantation; Reproductive Techniques; Thrombophilia
MeSH Terms: conditions — Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Both hereditary and acquired thrombophilia have been associated with recurrent miscarriage and pregnancy complications. Thrombophilia could favor the development of thrombosis of the maternal vasculature and obstacle placentation. Some studies have suggested a role of thrombophilia in the failure of assisted reproductive techniques although this association has been recently questioned. The scope of this study is to evaluate the effect of thrombophilia on the implantation rate and live birth rate in women undergoing ART.

Design: prospective, observational study Primary end-point: live birth rate. Secondary end-points: implantation rate, venous thromboembolic events during ART up to 6 weeks post-partum

ELIGIBILITY:
Inclusion Criteria:

* women undergoing ART
* age 18 years or older

Exclusion Criteria:

* ongoing anticoagulant therapy
* previous venous thromboembolism
* no informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women 18 years or older undergoing ART
Sampling Method: Non-Probability Sample
Enrollment: 687 (Actual)
Dates: Start 2015-01; Primary Completion 2017-07 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Live birth rate | Participants will be followed for the duration of the pregnancy, an expected average of 9 months

SECONDARY OUTCOMES:
implantation rate | Participants will be followed from the implantation to the ultrasonography to document the gestational sac, an expected average of 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Di Nisio, Principal Investigator — University G. D'Annunzio, Chieti, Italy
Locations (1):
- Universita degli Studi G. d'Annunzio Chieti e Pescara, Chieti, Italy